CLINICAL TRIAL: NCT00032084
Title: Smoking Cessation Intervention (Including Bupropion-Zyban Versus Placebo) for Completely Resected Stage I and II Non-Small Cell Lung Cancer Survivors Who Are Current Smokers
Brief Title: S0002 - A Program to Quit Smoking With or Without Bupropion in Treating Patients With Stage I or II Non-Small Cell Lung Cancer Who Have Undergone Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was closed early due to poor accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CDR0000069256; SWOG-S0002 (Other: SWOG); CALGB-79807 (Other: CALGB); ECOG-S0002 (Other: ECOG); NCI-P02-0215 (Other: NCI)
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Bupropion; Nicotine; Psychiatric Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral Intervention + Placebo (Placebo Comparator): Smoking cessation intervention , nicotine replacement, psychosocial assessment and care, and placebo.
  Interventions: Behavioral: smoking cessation intervention; Drug: nicotine; Procedure: psychosocial assessment and care
- Behavioral Intervention + Bupropion (Active Comparator): Smoking cessation intervention, nicotine replacement, psychosocial assessment and care, and bupropion hydrochloride .
  Interventions: Behavioral: smoking cessation intervention; Drug: bupropion hydrochloride; Drug: nicotine; Procedure: psychosocial assessment and care

INTERVENTIONS:
Behavioral: smoking cessation intervention — Physician will deliver the smoking cessation advice, reinforce the established quit date (no sooner than seven days after starting bupropion/placebo), and will distribute patient educational materials and all pharmacotherapy
Drug: bupropion hydrochloride — 150 mg/day on Days 1-3, 300 mg/day on Day 4-77
  Other Names: Zyban
  Arms: Behavioral Intervention + Bupropion
Drug: nicotine — 21 mg patch/day for Weeks 2-7; 14 mg patch/day for Weeks 8-9; 7 mg patch/day for Weeks 10-11.
  Other Names: Nicoderm CQ
Procedure: psychosocial assessment and care — The nurse/CRA will debrief the patients after the brief physician intervention and will follow-up with a series of 5 phone calls to provide booster advice. All advice will be based on the stage of change model (i.e., tailored to the patient's readiness to quit and/or stay off cigarettes).

SUMMARY:
RATIONALE: A program that includes bupropion may be more effective in helping early-stage lung cancer patients to quit smoking. It is not yet known if a program to quit smoking is more effective with or without bupropion.

PURPOSE: Randomized phase III trial to determine the effectiveness of a program to quit smoking with or without bupropion in treating patients who have undergone surgery for stage I or stage II non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of a smoking cessation intervention comprising behavior intervention and nicotine replacement with or without bupropion on 12-month quit rates in patients with completely resected stage I or II non-small cell lung cancer who are current smokers.
* Compare the predictors of smoking cessation success in patients treated with these regimens.
* Determine the relationship between smoking cessation and standard outcome measures (e.g., second malignancies, survival, and symptom status) in patients treated with these regimens.
* Compare the effect of these treatment regimens on emotional functioning in these patients.

OUTLINE: This is a randomized, double-blind, multicenter study. Patients are stratified according to gender, prior neoadjuvant or concurrent adjuvant chemotherapy and/or radiotherapy (yes vs no), and time since prior surgery (less than 6 months vs 6 to 12 months vs more than 12 months). Patients are randomized to 1 of 2 arms.

All patients receive behavioral intervention comprising smoking cessation advice and education on day 1. Patients quit smoking on day 8. Patients then receive a nicotine transdermal patch once daily on days 8-77.

* Arm I: Patients receive oral bupropion once daily on days 1-3 and twice daily on days 4-77.
* Arm II: Patients receive oral placebo as in arm I. Patients are followed at 3, 6, and 12 months and then annually for 10 years.

PROJECTED ACCRUAL: A total of 468 patients (234 [117 men and 117 women] per arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage I or II non-small cell lung cancer with complete resection of all disease

  * Must be free of recurrent or progressive disease
* Current smoker defined as:

  * Smoked at least 100 cigarettes in entire life AND
  * Currently smoking some days or every day
* Must establish a quit date that falls within 30 days after registration, but 7 days after physician advice and start of bupropion or placebo therapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* Not within an immediate post-infarction period
* No uncontrolled arrhythmias
* No unstable angina
* No uncontrolled hypertension (unstable blood pressure, diastolic pressure 90 mm Hg or greater)

Other:

* Must be able to read, speak, and understand English
* Must be willing to allow testing of saliva for cotinine levels
* No history of seizures
* No history of eating disorders
* No known drug-drug interactions between nicotine patch and/or bupropion and patient's current or planned medications including chemotherapy and antiemetics
* No concurrent psychiatric diagnosis that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Concurrent adjuvant chemotherapy allowed

Endocrine therapy:

* No concurrent systemic steroids

Radiotherapy:

* Concurrent adjuvant radiotherapy allowed

Surgery:

* See Disease Characteristics
* Recovered from prior surgery

Other:

* Prior neoadjuvant therapy allowed
* At least 14 days since prior medications containing bupropion (e.g., Wellbutrin or Wellbutrin SR)
* No other concurrent medications that contain bupropion (e.g., Wellbutrin or Wellbutrin SR)
* No concurrent monoamine oxidase inhibitors
* No concurrent medications that lower seizure threshold (e.g., antipsychotics, antidepressants, or theophylline)
* No other concurrent nicotine replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2002-01; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
To compare the effect on 12 month quit rates of adding an anti-depressant versus placebo in a double blind to an intervention and nicotine replacement in complete resected Stage I and II non-small cell lung cancer patients who are current smokers | 12 months

SECONDARY OUTCOMES:
To assess predictors of successful cessation in male and female patients. | 12 months
To explore the relationship between smoking cessation and standard outcome measures. | 12 months
To compare the effect on emotional functioning of adding bupropion to a behavioral intervention plus nicotine replacement in this patient population. | 12 months

OTHER OUTCOMES:
To explore the relationship of nicotine dependence genetic markers to 12 month quit rates by way of the dopamine D2 receptor gene (DRD2). | 12 months
To assess the relationship among metabolic polymorphism genes associated with lung cancer susceptibility in smokers who are lung cancer patients. | 12 months
To examine the relationship of nicotine susceptibility markers to 1 month quit rate, gender and pharmacologic (nicotine replacement therapy and either placebo or bupropion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ellen R. Gritz, PhD, Study Chair — M.D. Anderson Cancer Center; Philip C. Hoffman, MD, Study Chair — University of Chicago; James Stevenson, MD, Study Chair — Presbyterian medical center
Locations (176):
- United States (175):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center of Georgetown University Medical Center, Washington D.C., District of Columbia
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Hospital Comprehensive Cancer Center, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Saint Anthony Medical Center, Rockford, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Kansas Cancer Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Lakeland Medical Center - St. Joseph, Saint Joseph, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth Medical School, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - NorthEast Oncology Associates, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Lenoir Memorial Hospital Cancer Center, Kinston, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Danville Radiation Therapy Center, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - St. Mary's Medical Center, Huntington, West Virginia
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Ministry Medical Group - Northern Region, Rhinelander, Wisconsin
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico